CLINICAL TRIAL: NCT05785208
Title: Efficacy Study of Osimertinib in Treatment-naïve Patients With EGFR Mutant NSCLC According to TP53 Mutational Status.
Acronym: TEMPLE-2
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Bria Emilio, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4273
Record Dates: First submitted 2023-03-14; First posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Non Small Cell Lung Cancer
Keywords: TP53; EGFR; NSCLC; Osimertinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARM A: TP53 wilde-type (Experimental): Participants will receive osimertinib 80 mg once daily until disease progression or unacceptable toxicity.
  Interventions: Drug: Osimertinib
- ARM B: TP53 mutant (Experimental): Participants will receive osimertinib 80 mg once daily until disease progression or unacceptable toxicity.
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: Osimertinib — Osimertinib will be administered at a dose of 80 mg daily until disease progression

SUMMARY:
This is a prospective, biomarker-driven, open-label, clinical trial of osimertinib in treatment- naïve patients with EGFR mutant NSCLC, to evaluate the efficacy of osimertinib according to the TP53 mutational status.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures.
* Patients (male/female) must be > 18 years of age.
* Locally advanced or metastatic EGFR mutant NSCLC, not amenable to curative surgery or radiotherapy with confirmation of the presence of EGFR exon 19 deletion or exon 21 p.L858R.
* Mandatory provision of an unstained, archived tumour tissue sample in a quantity sufficient to allow central analysis.
* Patients must be treatment-naïve for locally advanced or metastatic NSCLC and eligible to receive first-line treatment with osimertinib. Prior adjuvant and neo-adjuvant therapy is permitted (chemotherapy, radiotherapy) if at least 6 months has elapsed between the end of chemotherapy and enrolment.
* World Health Organization (WHO) performance status 0-2.
* Patients must have a life expectancy ≥ 12 weeks.
* Females should be using adequate contraceptive measures, should not be breastfeeding and must have a negative pregnancy test prior to start of dosing if of child- bearing potential or must have evidence of non-child-bearing potential by fulfilling one of the following criteria at screening:

  1. Post-menopausal defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments.
  2. Women under 50 years old would be consider postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with LH and FSH levels in the post-menopausal range for the institution.
  3. Documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.
* Male patients should be willing to use barrier contraception.
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* At least one lesion, not previously irradiated, that can be accurately measured at baseline as ≥ 10 mm in the longest diameter (except lymph nodes which must have short axis ≥ 15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) and which is suitable for accurate repeated measurements.

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to both sponsor staff and/or staff at the study site).
* Previous treatment with osimertinib or other drugs targeting EGFR.
* Treatment with an investigational drug within five half-lives of the compound or 3 months, whichever is greater.
* Patients currently receiving (or unable to adequately stop use prior to receiving the first dose of study treatment) medications or herbal supplements included in Annex 6 (Guidance Regarding Potential Interactions with Concomitant Medications).
* Any unresolved toxicities from prior therapy greater than CTCAE grade 1 at the time of starting study treatment with the exception of alopecia and grade 2, prior platinum-therapy related neuropathy.
* Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension and active bleeding diatheses, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardise compliance with the protocol, or active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV). Screening for chronic conditions is not required.
* Patients with spinal cord compression, symptomatic and unstable brain metastases except for those patients who have completed definitive therapy, and have had a stable neurological status for at least 2 weeks after completion of definitive therapy. Patients may be on corticosteroids to control brain metastases if they have been on a stable dose for 2 weeks (14 days) prior to the start of study treatment and are clinically asymptomatic.
* Past medical history of ILD, drug-induced ILD, radiation pneumonitis requiring steroid treatment, or any evidence of clinically active ILD.
* Inadequate bone marrow reserve or organ function as demonstrated by any of the following laboratory values:

  1. Absolute neutrophil count <1.5 x 109/L.
  2. Platelet count <100 x 109/L.
  3. Haemoglobin <90 g/L.
  4. Alanine aminotransferase >2.5 times the upper limit of normal (ULN) if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases.
  5. Aspartate aminotransferase >2.5 times ULN if no demonstrable liver metastases or >5 times ULN in the presence of liver metastases.
  6. Total bilirubin >1.5 times ULN if no liver metastases or >3 times ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinemia) or liver metastases.
  7. Creatinine >1.5 times ULN concurrent with creatinine clearance <50 ml/min (measured or calculated by Cockcroft and Gault equation); confirmation of creatinine clearance is only required when creatinine is >1.5 times ULN.
* Any of the following cardiac criteria:

  1. Mean resting corrected QT interval (QTc using Fredericia's formula) > 470 msec.
  2. Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g., complete left bundle branch block, third degree heart block, and second degree heart block).
  3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, electrolyte abnormalities (including serum/plasma potassium < LLN, serum/plasma magnesium < LLN, and serum/plasma calcium <LLN), congenital long QT syndrome, family history of long QT syndrome or unexplained sudden death under 40 years of age in first degree relatives or any
* Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of osimertinib.
* Active second malignancy; i.e., patient known to have potentially fatal cancer present for which he/she may be (but not necessarily) currently receiving treatment. Patients with a history of malignancy that has been completely treated, with no evidence of that cancer currently, are permitted to enrol in the trial provided all chemotherapy was completed > 6 months prior and/or bone marrow transplant > 2 years prior to first day of study treatment.
* Patients with other serious diseases or clinical conditions, including but not limited to uncontrolled active infection and any other serious underlying medical processes that could affect the patient's capacity to participate in the study.
* History of hypersensitivity to osimertinib (or drugs with a similar chemical structure or class to osimertinib) or any excipients of these agents.
* Males and females of reproductive potential who are not using an effective method of birth control and females who are pregnant or breastfeeding or have a positive (urine or serum) pregnancy test prior to study entry.
* Judgment by the Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2022-06-28 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) According to RECIST v1.1 | 24 months
  PFS is defined as the time from randomization until the date of objective disease progression using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or death (by any cause) in the absence of progression, whichever comes first.

SECONDARY OUTCOMES:
Overall Survival (OS) | 24 months
  Overall Survival is defined as the time from the date of randomization to the date of participant's death due to any cause.
Objective Response Rate (ORR) | 24 months
  ORR is defined as the percentage of participants who achieve either a complete response (CR) or partial response (PR) using RECIST v1.1 criteria.
Disease Control Rate (DCR) | 24 months
  DCR is define as the percentage of patients who achieve complete response (CR), partial response (PR) or stable disease (SD)
Duration of Response (DoR) | 24 months
  DoR is defined as the time from the date of first documented response (CR or PR) until the date of documented progression or death, whichever comes first, only for participants who achieve CR or PR using RECIST v1.1 criteria.
Incidence and Severity of Adverse Events (AEs) according to CTCAE V5.0 | 24 months
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Time to Central Nervous System (CNS) progression | 24 months
  Time to CNS progression is defined as the time from randomization until the date of objective disease progression in the CNS using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
Objective Response Rate (ORR) in the Central Nervous System (CNS) | 24 months
  ORR in the CNS is defined as the percentage of participants who achieve either a complete response (CR) or partial response (PR) for CNS lesions using RECIST v1.1 criteria.

CONTACTS AND LOCATIONS:
Locations (11):
- Italy (11):
  - Azienda Ospedaliero-Universitaria Ospedali Riuniti, Ancona
  - IRCCS Istituto Tumori Giovanni Paolo II, Bari
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Ospedale Universitario di Parma, Parma
  - Ospedale San Camillo de Lellis, Rieti
  - Università Policlinico Tor Vergata, Rome
  - Policlinico Umberto I, Rome
  - Fondazione Policlinico Gemelli IRCCS, Rome
  - Ospedale San Giovanni-Addolorata, Rome
  - Ospedale San Luigi, Turin
  - Università degli Studi di Verona, Verona

IPD SHARING:
Plan to Share IPD: No